CLINICAL TRIAL: NCT06618690
Title: Efficacy of a Supervised Exercise Program on Pain, Physical Function, and Quality of Life in Breast Cancer Survivors: Protocol for a Randomized Clinical Trial
Brief Title: Exercise Program on Pain, Physical Function, and Quality of Life in Breast Cancer Survivors
Acronym: IO/2024
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IO/2024; IO/2024 (Other: Universidad de Burgos)
Record Dates: First submitted 2024-09-16; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Female Breast Cancer
Keywords: breast cancer; exercise; quality of life; muscle strength
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Grupo experimental (Experimental): The participants will be recruited through the oncologists of the Hospital Universitario Torrecárdenas (Almería). The proposal will be carried out in the intervention group (group 1), while the control group (group 2) will undergo the conventional recommendations indicated for this type of patients.
  Interventions: Other: Exercise program
- group control (No Intervention): The participants will be recruited through the oncologists of the Hospital Universitario Torrecárdenas (Almería). The proposal will be carried out in the intervention group (group 1), while the control group (group 2) will undergo the conventional recommendations indicated for this type of patients.

INTERVENTIONS:
Other: Exercise program — A supervised training plan will be carried out for 12 weeks with a frequency of 3 sessions per week with a duration of 60 minutes, an ideal estimate according to the meta-analysis of Montaño-Rojas et al. The first two weeks the group exercises will be performed to familiarize the participants with the exercises and then each participant will perform them at home with a review every two weeks to assess the increase of the load.
  The exercises and loads included in this treatment plan have been designed and modified based on previous clinical trials. The training plan will work upper limbs, lower limbs and trunk. All sessions begin with a general warm-up, which will be previously instructed to the participants, in which the heart rate will be increased (see Multimedia Appendix 1). After a two-minute break, the specific block of each session will begin (see Table 1 and Multimedia Appendix 1). All exercises will be performed with dumbbells, elastic bands and a ball.
  Arms: Grupo experimental

SUMMARY:
The purpose of this project is to develop a randomized clinical trial to determine the efficacy of a supervised exercise program on pain, physical function and quality of life in female breast cancer survivors

DETAILED DESCRIPTION:
A randomized, double-blind, clinical trial will be conducted with 325 participants. The intervention group will receive a supervised exercise program for 12 weeks, while the control group will receive no intervention. Participants' pain, physical function and quality of life will be assessed at baseline, post-intervention and 12 weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 65 years of age,
* women with oncologic treatment completed less than 3 months ago,
* women without metastasis,
* women without pathologies that contraindicate exercise,
* women who have agreed to sign the informed consent form

Exclusion Criteria:

* not attending scheduled sessions to instruct on the exercises to be performed, - being part of other studies,
* undergoing another type of therapy
* pregnancy patients.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
repeated measures ANOVA | 12 weeks
  the range of motion, tone and muscle strength of the group will be measured in 3 measures over the 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Torrecárdenas, Àlmeria, Alemeria, Spain

IPD SHARING:
Plan to Share IPD: No
A randomized, double-blind, clinical trial will be conducted with 325 participants. The intervention group will receive a supervised exercise program for 12 weeks, while the control group will receive no intervention. Participants' pain, physical function and quality of life will be assessed at baseline, post-intervention and 12 weeks post-intervention.

REFERENCES:
- [Background] Iwase T, Wang X, Shrimanker TV, Kolonin MG, Ueno NT. Body composition and breast cancer risk and treatment: mechanisms and impact. Breast Cancer Res Treat. 2021 Apr;186(2):273-283. doi: 10.1007/s10549-020-06092-5. Epub 2021 Jan 21. PMID 33475878
- [Background] Michels D, Konig S, Heckel A. Effects of combined exercises on shoulder mobility and strength of the upper extremities in breast cancer rehabilitation: a 3-week randomized controlled trial. Support Care Cancer. 2023 Sep 1;31(9):550. doi: 10.1007/s00520-023-07959-1. PMID 37656241
- [Background] Tuchler A, De Pauw A, Ernst C, Anota A, Lakeman IMM, Dick J, van der Stoep N, van Asperen CJ, Maringa M, Herold N, Blumcke B, Remy R, Westerhoff A, Stommel-Jenner DJ, Frouin E, Richters L, Golmard L, Kutting N, Colas C, Wappenschmidt B, Rhiem K, Devilee P, Stoppa-Lyonnet D, Schmutzler RK, Hahnen E. Clinical implications of incorporating genetic and non-genetic risk factors in CanRisk-based breast cancer risk prediction. Breast. 2024 Feb;73:103615. doi: 10.1016/j.breast.2023.103615. Epub 2023 Nov 29. PMID 38061307
- [Derived] Garcia-Molina J, Saiz-Vazquez O, Santamaria-Vazquez M, Ortiz-Huerta JH. Efficacy of a Supervised Exercise Program on Pain, Physical Function, and Quality of Life in Patients With Breast Cancer: Protocol for a Randomized Clinical Trial. JMIR Res Protoc. 2025 Mar 12;14:e63891. doi: 10.2196/63891. PMID 40073395